CLINICAL TRIAL: NCT02239744
Title: Cardiopulmonary Benefits of Reducing Indoor Particles of Outdoor Origin: a Randomized Double-blind Crossover Trial of Air Purifiers
Brief Title: Intervention Study on the Health Impact of Air Filters in Chinese Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Haidong Kan, PhD and Professor, Fudan University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: FDUEH-1
Record Dates: First submitted 2014-09-07; First posted 2014-09-15 (Estimated); Results first posted 2014-12-01 (Estimated); Last update posted 2016-01-13 (Estimated); Status verified 2016-01

CONDITIONS: Inflammation; Coagulation; Blood Pressure; Pulmonary Function
Keywords: air pollution; air purification; intervention; randomized controlled trial; cardiovascular health; pulmonary health
MeSH Terms: conditions — Inflammation; Thrombosis | interventions — Air Filters

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- True air purification (Experimental): One group of subjects used an intervention of true air purifiers placed in the center of the room.
  Interventions: Behavioral: Air purifiers
- Sham air purification (Sham Comparator): This group of subjects used an intervention of sham air purifiers under the same conditions with true purifiers with the only difference being removal of the filter gauze in the sham purifiers.
  Interventions: Behavioral: Air purifiers

INTERVENTIONS:
Behavioral: Air purifiers — The 10 dormitory rooms were randomized into two groups of 5 rooms each. One group used an air purifier placed in the center of the room for 48 hours corresponding to one weekend, followed by a 2-week washout period, and another 48 hours of using a sham air purifier under the same conditions. The other group simply reversed the order in which the real and sham air purifiers were used. All rooms used the same qualified air purifiers (model FAP04, 3M Filtrete), with the only difference being removal of the filter gauze in the sham purifiers. The air pollution auto-sensing feature of air purifiers was disabled in both groups. All participants and research staff were blinded to the group assignment. We requested all participants to stay in their dormitory room with the windows/doors closed throughout each 48-hour intervention period.
  Other Names: Air filtration

SUMMARY:
This study aimed to evaluate whether a short-term indoor air purifier intervention improves cardiopulmonary health based on a randomized double-blind crossover trial

DETAILED DESCRIPTION:
We conducted a randomized double-blind crossover trial among 35 healthy college students in Shanghai, China in 2014. These students lived in dormitories that were randomized into two groups and alternated the use of true or sham air purifiers for 48 hours with a 2-week wash-out interval.All participants and research staff were blinded to the group assignment. We requested all participants to stay in their dormitory room with the windows/doors closed throughout each 48-hour intervention period. We delivered foods and drinks to each room during the intervention period. All interventions started at 8 a.m. to avoid issues related to diurnal variation. We evaluated health endpoints and drew blood immediately after the completion of each 48-hour intervention. We measured 14 circulating biomarkers of inflammation, coagulation and vasoconstriction, lung function, blood pressure (BP), and fractional exhaled nitric oxide (FeNO).

ELIGIBILITY:
Inclusion Criteria:

* Healthy college students aged between 18 and 26
* All the subjects should stay indoor almost the entire time, and stayed within the central urban area of shanghai during the wash-out period.

Exclusion Criteria:

* current smokers or ever smokers
* chronic respiratory diseases
* chronic cardiovascular diseases
* acute infections
* medication use in recent one month

Ages: 18 Years to 26 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2014-09; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Haidong Kan, PhD, Study Director — School of Public Health，Fudan University
Locations (1):
- Department of Environmental Health, School of Public Health, Fudan University, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Chen R, Zhao A, Chen H, Zhao Z, Cai J, Wang C, Yang C, Li H, Xu X, Ha S, Li T, Kan H. Cardiopulmonary benefits of reducing indoor particles of outdoor origin: a randomized, double-blind crossover trial of air purifiers. J Am Coll Cardiol. 2015 Jun 2;65(21):2279-87. doi: 10.1016/j.jacc.2015.03.553. PMID 26022815

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We recruited 35 healthy college students.
Pre-assignment Details: We recruited 35 healthy college students and no one were excluded according to the exclusion criteria.
Groups:
- Sham Purifiers First, Then True Purifiers: The 10 rooms were randomized into two groups of 5 rooms each. In the first period, this group used sham air purifiers with the only difference being removal of the filter gauze. In the second period, this group used true air purifiers.
- True Purifiers First, Then Sham Purifiers: The 10 rooms were randomized into two groups of 5 rooms each. In the first period, this group used true air purifiers.In the second period, this group used sham air purifiers.
Period: Period 1
Arm/Group | Sham Purifiers First, Then True Purifiers | True Purifiers First, Then Sham Purifiers
Started | 17 | 18
Completed | 17 | 18
Not Completed | 0 | 0
Period: Period 2
Arm/Group | Sham Purifiers First, Then True Purifiers | True Purifiers First, Then Sham Purifiers
Started | 17 | 18
Completed | 17 | 18
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All 35 participants recivered palecbo and real intervention, and the order was random. This crossover study autonomically allows each subject to serve as his or her own control over time.
Groups:
- Sham Purifiers: The 10 rooms were randomized into two groups of 5 rooms each. This group used sham air purifiers with the only difference being removal of the filter gauze.
- True Purifiers: The 10 rooms were randomized into two groups of 5 rooms each. This group used true air purifiers.
- Total: Total of all reporting groups
Arm/Group | Sham Purifiers | True Purifiers | Total
Number analyzed (Participants) | 17 | 18 | 35
Age, Continuous [Mean (Standard Deviation); unit: years] — We recruited all participants from the Fenglin campus of Fudan University. Therefore, all these students are young adult whose age was nearly 23 years old.
  years | 24 (2) | 21 (2) | 23 (2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 13 | 25
  Male | 5 | 5 | 10
Region of Enrollment [Number; unit: participants]
  China | 17 | 18 | 35
BMI [Mean (Standard Deviation); unit: Kg/m^2] | 21 (2.5) | 22 (2.5) | 22 (2.5)

OUTCOME MEASURES:

1. Primary Outcome: Circulating Biomarkers
Description: Peripheral blood samples (5 ml) were drawn by a nurse, separated into serum and plasma, and stored at -80 ℃ within 30 minutes. We measured the levels of 14 circulating biomarkers: (1) 8 biomarkers of inflammation, including C-reactive protein (CRP), fibrinogen, P-selection, monocyte chemoattractant protein-1 (MCP-1), interleukin-1b, interleukin-6, tumor necrosis factor-α (TNF-α) and myeloperoxidase; (2) 4 biomarkers of coagulation, including soluble CD40 ligand (sCD40L), plasminogen activator inhibitor-1, tissue plasminogen activator and D-Dimer; and (3) 2 biomarkers of vasoconstriction, including endothelin-1 and angiotensin-converting enzyme.
Time Frame: Blood samples were drawn within one hour after the intervention, and lab analysis was completed in the next 10 days
Measure: Geometric Mean (Standard Deviation); unit: ng/ml
Arm/Group | Sham Purifiers | True Purifiers
Number analyzed (Participants) | 35 | 35
ng/ml
  C-reaction protein（CRP） | 926.3 (1967.1) | 913.1 (1734.0)
  Fibrinogen | 1122.2 (280.1) | 1108.2 (232.8)
  P-selection | 139.0 (41.6) | 129.4 (39.3)
  Soluble CD40L ligand（sCD40L） | 1.4 (1.6) | 0.5 (1.1)
  plasminogen activator inhibitor-1（PAI-1） | 54.9 (16.7) | 41.5 (20.0)
  Myeloperoxidase（MPO） | 1579.4 (772.0) | 1261.4 (659.4)
  D-Dimer | 1174.6 (817.2) | 1001.2 (988.5)
  Angiotensin-converting enzyme（ACE） | 102.9 (32.4) | 101.1 (31.9)

2. Secondary Outcome: Blood Pressure
Description: After sitting in a quiet room for at least 5 min, participants had their left upper arm BP measured by trained technicians using a mercury sphygmomanometer at least three times with 2-min minimum intervals between measurements. The second and third sets of readings were averaged to obtain systolic BP and diastolic BP. Pulse pressure was calculated as the difference between systolic BP and diastolic BP. If the differences among the three measurements were bigger than 5 mmHg, a new round of measurements were arranged.
Time Frame: Within one hour after the 2-day intervention
Measure: Geometric Mean (Standard Deviation); unit: mmHg
Arm/Group | Sham Purifiers | True Purifiers
Number analyzed (Participants) | 35 | 35
mmHg
  Systolic pressure | 106.0 (9.6) | 103.0 (10.2)
  Diastolic pressure | 70.9 (8.6) | 67.9 (8.9)
  Pulse pressure | 34.8 (5.4) | 34.8 (5.9)

3. Primary Outcome: Lung Function
Description: A respiratory physician measured forced vital capacity, forced expiratory volume in 1 second and peak expiratory flow of each participant using the JAEGER Masterlab equipment (Würzburg, Germany) that meets the American Thoracic Society criteria. The volume signal was calibrated at least once on a testing day with a 3.0 L syringe connected to the pneumotachograph in accordance with the manufacturers' recommendations. We instructed participants to perform at least three forced expiratory lung function maneuvers in order to obtain a minimum of two acceptable and reproducible values, and we recorded the best results.
Time Frame: Within 1 hour after the end of the two-day intervention
Population: Ultimately, all 35 participants completed this study.This crossover study autonomically allows each subject to serve as his or her own control over time.
Measure: Geometric Mean (Standard Deviation); unit: L
Arm/Group | Sham Purifiers | True Purifiers
Number analyzed (Participants) | 35 | 35
L
  forced vital capacity(FVC) | 3.0 (0.7) | 3.1 (0.8)
  forced expiratory volume in 1 s(FEV1) | 2.8 (0.5) | 2.8 (0.5)

4. Secondary Outcome: Fractional Exhaled Nitric Oxide
Description: FeNO is an established biomarker of respiratory inflammation, and has been widely used in epidemiological studies because of its high sensitivity, specificity and non-invasive nature. We measured FeNO levels using a portable NIOX MINO machine (Aerocrine AB, Solna, Sweden) according to standardized procedures by the American Thoracic Society and the European Respiratory Society.
Time Frame: within 1 hour after the two-day intervention
Measure: Geometric Mean (Standard Deviation); unit: ppb
Arm/Group | Sham Purifiers | True Purifiers
Number analyzed (Participants) | 35 | 35
ppb | 14.5 (25.1) | 13.3 (20.6)

ADVERSE EVENTS:
Time Frame: At the end of each 2-day period
Arm/Group | Sham Purifiers | True Purifiers
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/35
Other Adverse Events (participants affected / at risk) | 0/35 | 0/35

LIMITATIONS AND CAVEATS:
The study only included 35 participants in 10 rooms, we might therefore have missed some potentially important but modest differences due to the relatively small sample size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes